CLINICAL TRIAL: NCT00119366
Title: A Phase II Trial Combining Radiolabeled BC8 (Anti-CD45) Antibody With Fludarabine and Low Dose TBI Followed by Related or Unrelated PBSC Infusion and Post-Transplant Immunosuppression for Patients With Advanced AML or High Risk Myelodysplastic Syndrome
Brief Title: Iodine I 131 Monoclonal Antibody BC8, Fludarabine Phosphate, Total Body Irradiation, and Donor Stem Cell Transplant Followed by Cyclosporine and Mycophenolate Mofetil in Treating Patients With Advanced Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ended before target accrual was reached; participants are no longer being examined or receiving intervention.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Johnnie Orozco, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1809.00; NCI-2010-00234 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1809.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2005-07-12; First posted 2005-07-13 (Estimated); Results first posted 2022-08-01 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Childhood Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Refractory Anemia With Ringed Sideroblasts; Refractory Cytopenia With Multilineage Dysplasia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — fludarabine phosphate; Whole-Body Irradiation; Peripheral Blood Stem Cell Transplantation; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Intervention Model Description: This study will assess the feasibility and safety of patients with advanced AML or high-risk MDS treated with Iodine-131 BC8 antibody at a starting dose of 22 Gy delivered to the normal organ receiving the highest dose combined with fludarabine and 2 Gy total body irradiation (TBI), plus cyclosporine (CSP)/mycophenolate mofetil (MMF), followed by matched related or unrelated allogeneic hematopoietic stem cell transplantation (HSCT). Determination of the maximum tolerated dose (MTD) will be the major study endpoint.
  Dose-escalation/de-escalation of radiolabeled BC8 antibody (I-131-BC8) is conducted using a "two-stage" approach. Under this plan, dose levels during the first stage are increased (or decreased) for individual patients until a dose-limiting toxicity (DLT) is observed, at which point the second stage proceeds with each dose level administered to a cohort of four patients.
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose Level 1: 12 Gy iodine-131 monoclonal antibody BC8 (Experimental): RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  Interventions: Radiation: iodine I 131 monoclonal antibody BC8; Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis
- Dose Level 7: 22 Gy iodine-131 monoclonal antibody BC8 (Experimental): RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  Interventions: Radiation: iodine I 131 monoclonal antibody BC8; Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis
- Dose Level 8: 24 Gy iodine-131 monoclonal antibody BC8 (Experimental): RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  Interventions: Radiation: iodine I 131 monoclonal antibody BC8; Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis
- Dose Level 9: 26 Gy iodine-131 monoclonal antibody BC8 (Experimental): RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  Interventions: Radiation: iodine I 131 monoclonal antibody BC8; Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis
- Dose Level 10: 28 Gy iodine-131 monoclonal antibody BC8 (Experimental): RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  Interventions: Radiation: iodine I 131 monoclonal antibody BC8; Drug: fludarabine phosphate; Radiation: total-body irradiation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis

INTERVENTIONS:
Radiation: iodine I 131 monoclonal antibody BC8 — Given IV
  Other Names: I 131 MOAB BC8; I 131 Monoclonal Antibody BC8; iodine I 131 MOAB BC8
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo PBSC transplantation
Procedure: peripheral blood stem cell transplantation — Undergo PBSC transplantation
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Drug: cyclosporine — Given IV or PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; MMF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and best dose of iodine I 131 monoclonal antibody BC8 when given together with fludarabine phosphate, total-body irradiation, and donor stem cell transplant followed by cyclosporine and mycophenolate mofetil in treating patients with acute myeloid leukemia or myelodysplastic syndrome that has spread to other places in the body and usually cannot be cured or controlled with treatment. Giving chemotherapy drugs, such as fludarabine phosphate, and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer or abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. Also, radiolabeled monoclonal antibodies, such as iodine I 131 monoclonal antibody BC8, can find cancer cells and carry cancer-killing substances to them without harming normal cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving fludarabine phosphate and total-body irradiation before the transplant together with cyclosporine and mycophenolate mofetil after the transplant may stop this from happening. Giving a radiolabeled monoclonal antibody together with donor stem cell transplant, cyclosporine, and mycophenolate mofetil may be an effective treatment for advanced acute myeloid leukemia or myelodysplastic syndromes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the maximum tolerated dose (MTD) and the transplant-related mortality (TRM) and toxicity of delivering 131I-BC8 (iodine I 131 monoclonal antibody BC8) (anti-cluster of differentiation [CD]45 antibody) at a starting dose of 22 Gy to the normal organ receiving the highest dose in combination with the non-myeloablative regimen of fludarabine (fludarabine phosphate) (FLU), 2 Gy total body irradiation (TBI), cyclosporine (CSP), mycophenolate mofetil (MMF), and human leukocyte antigen (HLA)-matched related or unrelated allogeneic hematopoietic stem cell transplant (HSCT) in patients 16 to 50 years old who have advanced acute myeloid leukemia (AML) or high risk myelodysplastic syndrome (MDS).

II. To estimate rates of donor chimerism resulting from this combined preparative regimen and to correlate level of donor chimerism with estimated radiation doses delivered to hematopoietic tissues via antibody.

III. To determine rates of disease relapse, graft vs. host disease, and 2-year disease-free survival in patients receiving 131I-BC8 antibody combined with FLU, 2 Gy TBI, CSP, MMF, and HLA-matched related or unrelated allogeneic HSCT.

OUTLINE: This is a dose-escalation study of iodine I 131 monoclonal antibody BC8.

RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 intravenously (IV) on day -12.

CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.

TRANSPLANTATION: After completion of TBI, patients undergo allogeneic peripheral blood stem cell (PBSC) transplant on day 0.

IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or orally (PO) twice daily (BID) on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO thrice daily (TID) on days 0 to 40 followed by a taper to day 96.

After completion of study treatment, patients are followed up at 6, 9, 12, 18, and 24 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced AML defined as beyond first remission, primary refractory disease, or evolved from myelodysplastic or myeloproliferative syndromes; or patients with MDS expressed as refractory anemia with excess blasts (RAEB), refractory anemia with excess blasts in transformation (RAEBT), refractory cytopenia with multilineage dysplasia (RCMD), RCMD with ringed sideroblasts (RCMD-RS), or chronic myelomonocytic leukemia (CMML)
* Patients not in remission must have CD45-expressing leukemic blasts or myelodysplastic cells; patients in remission do not require phenotyping and may have leukemia previously documented to be CD45 negative (because in remission patients, virtually all antibody binding is to non-malignant cells which make up >= 95% of nucleated cells in the marrow)
* Patients should have a circulating blast count of less than 10,000/mm^3 (control with hydroxyurea or similar agent is allowed)
* Patients must have an estimated creatinine clearance greater than 50/ml per minute (serum creatinine value must be within 28 days prior to registration)
* Bilirubin < 2 times the upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2 times the upper limit of normal
* Karnofsky score >= 70 or Eastern Cooperative Oncology Group (ECOG) =< 2
* Patients must have an expected survival of > 60 days and must be free of active infection
* Patients must have an HLA-identical sibling donor or an HLA-matched unrelated donor who meets standard Seattle Cancer Care Alliance (SCCA) and/or National Marrow Donor Program (NMDP) or other donor center criteria for peripheral blood stem cell (PBSC) donation; related donors should be matched by molecular methods at the intermediate resolution level at HLA-A, B, C, and developmentally regulated RNA binding protein 1 (DRB1) according to Fred Hutchinson Cancer Research Center (FHCRC) Standard Practice Guidelines and to the allele level at DQB1; unrelated donors should be identified using matching criteria that follows the FHCRC Standard Practice Guidelines limiting the study to eligible donors that are allele matched for HLA-A, B, C, DRB1, and DQB1 (grade 1), and accepting up to one allele mismatch as per Standard Practice grade 2.1 for HLA-A, B, or C
* DONOR: Donors must meet HLA matching criteria as well as standard SCCA and/or NMDP or other donor center criteria for PBSC donation

Exclusion Criteria:

* Circulating antibody against mouse immunoglobulin (human anti-mouse antibody [HAMA])
* Prior radiation to maximally tolerated levels to any normal organ
* Patients may not have symptomatic coronary artery disease and may not be on cardiac medications for anti-arrhythmic or inotropic effects
* Inability to understand or give an informed consent
* Patients who are seropositive for human immunodeficiency virus (HIV)
* Perceived inability to tolerate diagnostic or therapeutic procedures, particularly treatment in radiation isolation
* Patients who have previously undergone autologous or allogeneic HSCT

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2003-05; Primary Completion 2014-08 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnnie Orozco, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighteen participants enrolled in the study:
  16 - received & completed study treatment
  02 - withdrawn from the study
Pre-assignment Details: Dose escalation plan: single patients will be entered on the first stage, and escalation by 2 Gy increments in the radiation dose delivered to the normal organ receiving the highest dose will occur until a patient experiences a Grade III/IV regimen-related toxicity (Bearman) or dose-limiting toxicity (DLT), at which point the second stage will begin at the next lower dose level. If the first patient (i.e., at the starting dose level) has DLT, de-escalation will occur by 2 Gy increments
Groups:
- Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 7: 22 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 8: 24 Gy Iodine-131+ BC8 Monoclonal Antibody; Dose Level 9: 26 Gy Iodine-131+ BC8 Monoclonal Antibody; Dose Level 10: 28 Gy Iodine-131+ BC8 Monoclonal Antibody: RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  iodine I 131 monoclonal antibody BC8: Given IV
  fludarabine phosphate: Given IV
  total-body irradiation: Undergo TBI
  allogeneic hematopoietic stem cell transplantation: Undergo PBSC transplantation
  peripheral blood stem cell transplantation: Undergo PBSC transplantation
  cyclosporine: Given IV or PO
  mycophenolate mofetil: Given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 24 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 9: 26 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 10: 28 Gy Iodine-131+ BC8 Monoclonal Antibody
Started | 1 | 2 | 3 | 2 | 8
Completed | 1 | 2 | 3 | 2 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 8: 24 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 9: 26 Gy Iodine-131 + BC8 Monoclonal Antibody; Dose Level 10: 28 Gy Iodine-131 + BC8 Monoclonal Antibody: RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  iodine I 131 monoclonal antibody BC8: Given IV
  fludarabine phosphate: Given IV
  total-body irradiation: Undergo TBI
  allogeneic hematopoietic stem cell transplantation: Undergo PBSC transplantation
  peripheral blood stem cell transplantation: Undergo PBSC transplantation
  cyclosporine: Given IV or PO
  mycophenolate mofetil: Given PO
  laboratory biomarker analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 9: 26 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 10: 28 Gy Iodine-131 + BC8 Monoclonal Antibody | Total
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3 | 2 | 8 | 16
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 1 | 4 | 7
  Male | 0 | 2 | 2 | 1 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 2 | 2 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 2 | 2 | 2 | 7 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3 | 2 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT) 100 Days After Transplant
Description: The criteria of Grade III/IV regimen-related toxicity (Bearman) or dose-limiting toxicity (DLT) are as follows:
  Grade 1 Development of transient chemical abnormalities which are not of major clinical consequence and which reverse without requiring major medical interventions. In general, the intent of this toxicity scale is to observe transient target organ toxicity which is reversible.
  Grade 2 Development of chemical or laboratory abnormalities that are persistent and which may represent target organ damage that may not be readily reversed. It is anticipated that at this dose of the drug, the toxicity obtained would be manageable by clinical methods but may interfere with other therapies.
  Grade 3 Development of major clinical, chemical or laboratory abnormalities which represent maximum toxicities without being fatal. This grade of toxicity is designed to be the dose-limiting toxicity.
Time Frame: Up to 100 days post-transplant
Population: Study participants that received and completed study treatment
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 8: 24 Gy Iodine-131 + BC8; Dose Level 9: 26 Gy Iodine-131 + BC8; Dose Level 10: 28 Gy Iodine-131 + BC8: RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  iodine I 131 monoclonal antibody BC8: Given IV
  fludarabine phosphate: Given IV
  total-body irradiation: Undergo TBI
  allogeneic hematopoietic stem cell transplantation: Undergo PBSC transplantation
  peripheral blood stem cell transplantation: Undergo PBSC transplantation
  cyclosporine: Given IV or PO
  mycophenolate mofetil: Given PO
  laboratory biomarker analysis: Correlative studies
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 24 Gy Iodine-131 + BC8 | Dose Level 9: 26 Gy Iodine-131 + BC8 | Dose Level 10: 28 Gy Iodine-131 + BC8
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
Participants
  Number of participants with no dose-limiting toxicities 100 days after transplant | 1 | 2 | 3 | 2 | 8
  Number of participants with dose-limiting toxicities 100 days after transplant | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Transplant Related Mortality Within 100 Days After Transplant
Description: Number of participants that received and completed study treatment who died within 100 days after transplant
Time Frame: Up to 100 days post-transplant
Population: Participants that received and completed study treatment who died within 100 days after transplant
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1: 12 Gy Iodine-131+ BC8 Monoclonal Antibody: RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  iodine I 131 monoclonal antibody BC8: Given IV
  fludarabine phosphate: Given IV
  total-body irradiation: Undergo TBI
  allogeneic hematopoietic stem cell transplantation: Undergo PBSC transplantation
  peripheral blood stem cell transplantation: Undergo PBSC transplantation
  cyclosporine: Given IV or PO
  mycophenolate mofetil: Given PO
  laboratory biomarker analysis: Correlative studies
- Dose Level 7: 22 Gy Iodine-131+ BC8 Monoclonal Antibody; Dose Level 8: 24 Gy Iodine-131+ BC8 Monoclonal Antibody; Dose Level 9: 26 Gy Iodine-131+ BC8 Monoclonal Antibody; Dose Level 10: 28 Gy Iodine-131+ BC8: RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  iodine I 131 monoclonal antibody BC8: Given IV
  fludarabine phosphate: Given IV
  total-body irradiation: Undergo TBI
  allogeneic hematopoietic stem cell transplantation: Undergo PBSC transplantation
  peripheral blood stem cell transplantation: Undergo PBSC transplantation
  cyclosporine: Given IV or PO
  mycophenolate mofetil: Given PO
  laboratory biomarker analysis: Correlative studie
Arm/Group | Dose Level 1: 12 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 7: 22 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 8: 24 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 9: 26 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 10: 28 Gy Iodine-131+ BC8
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
Participants
  Number of participants who died within 100 days after transplant | 1 | 0 | 0 | 0 | 1
  Number of participants who are alive > 100 days after transplant | 0 | 2 | 3 | 2 | 7

3. Secondary Outcome: Participant Disease Response Within 4 Weeks After Transplant
Description: The number of participants that are in complete remission (CR) or relapsed within 4 weeks after transplant.
  Complete Remission is defined as complete resolution of all signs of leukemia for at least four weeks with all of the following:
  * Normal bone marrow with blasts <5% with normal cellularity, normal megakarypoiesis, more than 15% erythropoiesis and more than 25% granulocytopoiesis.
  * Normalization of blood counts (no blasts, platelets >100,000/mm3, granulocytes >1,500/mm3).
  * No extramedullary disease.
  Relapse is measured as follows:
  * After CR: >5% blasts in the bone marrow and/or peripheral blood.
  * Confirmation of relapse by bone marrow analysis with more than 10% blasts.
  * Extramedullary disease confirmed cytologically or histologically.
Time Frame: 4 weeks after transplant
Population: Participants that received and completed study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 9: 26 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 10: 28 Gy Iodine-131 + BC8 Monoclonal Antibody
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
Participants
  Number of participants that are in CR 4 weeks after transplant | 0 | 2 | 3 | 1 | 6
  Number of participants that relapsed 4 weeks after transplant | 1 | 0 | 0 | 1 | 2

4. Secondary Outcome: Severity of Acute GVHD in Patients Who Completed the Study Treatment
Description: The severity of acute GVHD is measured based on Graft-vs-Host Disease:
  Severity of GVHD Grade I +1 to +2 skin rash No gut or liver involvement
  Grade II +3 skin rash or
  * 1 gastrointestinal involvement and/or +1 liver involvement
  Grade III +2 to +4 gastrointestinal involvement and/or
  * 2 to +4 liver involvement with or without a rash
  Grade IV Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: 100 days after transplant
Population: Study participants that completed study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 12 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 7: 22 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 8: 24 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 9: 26 Gy Iodine-131 + BC8 Monoclonal Antibody | Dose Level 10: 28 Gy Iodine-131 + BC8 Monoclonal Antibody
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
Participants
  Number of participants with Grade 0-1 GVHD | 0 | 0 | 0 | 0 | 3
  Number of participants with Grade 2 GVHD | 1 | 2 | 3 | 2 | 4
  Number of participants with Grade 3 GVHD | 0 | 0 | 0 | 0 | 1

5. Secondary Outcome: Number of Participants With 100% Donor Chimerism at Day 28 and Day 84
Description: Post-transplant bone marrow samples were collected on day 28 and day 84 after transplant for DNA Chimerism Analysis
Time Frame: Day 28 and Day 80 after transplant
Population: Patients that completed the study regimen
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 12 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 7: 22 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 8: 24 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 9: 26 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 10: 28 Gy Iodine-131+ BC8
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
Participants
  Day 28 Donor Chimerism | 0 | 1 | 3 | 2 | 7
  Day 84 Donor Chimerism | 0 | 1 | 3 | 2 | 4

6. Secondary Outcome: Two-year Disease-free Survival of Study Participants Who Completed the Study Regimen
Description: Survival and complete resolution of all signs of leukemia for 2 years after transplant with all of the following:
  1. Normal bone marrow with blasts <5% with normal cellularity, normal megakarypoiesis, more than 15% erythropoiesis and more than 25% granulocytopoiesis.
  2. Normalization of blood counts (no blasts, platelets >100,000/mm3, granulocytes >1,500/mm3).
  3. No extramedullary disease.
Time Frame: 2 years post transplant
Population: Participants who are alive and disease-free 2 years after transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 12 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 7: 22 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 8: 24 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 9: 26 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 10: 28 Gy Iodine-131+ BC8
Number analyzed (Participants) | 1 | 2 | 3 | 2 | 8
Participants | 0 | 2 | 1 | 0 | 2

ADVERSE EVENTS:
Time Frame: Serious adverse events and Other (not including serious adverse events) were monitored and recorded from the time of first exposure to the investigational product (i.e. Iodine 131 + BC8 mAB) through day +100 post-transplant or through patient discharge from the Seattle Cancer Care Alliance (SCCA) system to the patient's primary physician. All-Cause Mortality was monitored/assessed for up to 2 years or through participant survival after completing the study regimen and transplant.
Groups:
- Dose Level 7: 22 Gy Iodine-131+ BC8 Monoclonal Antibody; Dose Level 8: 24 Gy Iodine-131+ BC8 Monoclonal Antibody; Dose Level 9: 26 Gy Iodine-131+ BC8 Monoclonal Antibody; Dose Level 10: 28 Gy Iodine-131+ BC8 Monoclonal Antibody: RADIOIMMUNOTHERAPY: Patients receive therapeutic iodine I 131 monoclonal antibody BC8 IV on day -12.
  CONDITIONING: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: After completion of TBI, patients undergo allogeneic PBSC transplant on day 0.
  IMMUNOSUPPRESSION: Patients with a matched related donor receive cyclosporine IV or PO BID on days -3 to 56 followed by a taper to day 180 in the absence of graft-versus-host disease. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO 2 BID on days 0 to 27. Patients with a matched unrelated donor receive cyclosporine IV or PO BID on days -3 to 100 followed by a taper to day 180. Beginning 4-6 hours after PBSC transplant, these patients also receive mycophenolate mofetil PO TID on days 0 to 40 followed by a taper to day 96.
  iodine I 131 monoclonal antibody BC8: Given IV
  fludarabine phosphate: Given IV
  total-body irradiation: Undergo TBI
  allogeneic hematopoietic stem cell transplantation: Undergo PBSC transplantation
  peripheral blood stem cell transplantation: Undergo PBSC transplantation
  cyclosporine: Given IV or PO
  mycophenolate mofetil: Given PO
  laboratory biomarker analysis: Correlative studies
Arm/Group | Dose Level 1: 12 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 7: 22 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 8: 24 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 9: 26 Gy Iodine-131+ BC8 Monoclonal Antibody | Dose Level 10: 28 Gy Iodine-131+ BC8 Monoclonal Antibody
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/2 | 2/3 | 2/2 | 2/8
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 3/3 | 2/2 | 8/8
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 1/3 | 2/2 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 12 Gy Iodine-131+ BC8 Monoclonal Antibody (N=1) | Dose Level 7: 22 Gy Iodine-131+ BC8 Monoclonal Antibody (N=2) | Dose Level 8: 24 Gy Iodine-131+ BC8 Monoclonal Antibody (N=3) | Dose Level 9: 26 Gy Iodine-131+ BC8 Monoclonal Antibody (N=2) | Dose Level 10: 28 Gy Iodine-131+ BC8 Monoclonal Antibody (N=8)
Engraftment Syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Atrial Fibrillation
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) — Low blood pressure
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rigors/Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Difficulty swallowing
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 1 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2) — Neutropenic fever
Infection - Other (Pulmonary Aspirgillus) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection - Other (C. Difficile) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurology- Other (altered mental status) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extremity/Limb (Left shoulder) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Acute Respiratory Distress Syndrome
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: 12 Gy Iodine-131+ BC8 Monoclonal Antibody (N=1) | Dose Level 7: 22 Gy Iodine-131+ BC8 Monoclonal Antibody (N=2) | Dose Level 8: 24 Gy Iodine-131+ BC8 Monoclonal Antibody (N=3) | Dose Level 9: 26 Gy Iodine-131+ BC8 Monoclonal Antibody (N=2) | Dose Level 10: 28 Gy Iodine-131+ BC8 Monoclonal Antibody (N=8)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Allergic reaction/hypersensitivity (including drug fever)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) — Anorexia
Hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Hearing loss
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Leukocytes (total WBC)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Neutrophils/granulocytes (ANC/AGC)
Platelets (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Platelets
WBC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — WBC
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Hypertension
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pericardial effusion
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) — Fatigue
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Fever
Rigors/chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Rigors/chills
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Rash/desquamation
Hot flashes/flushes (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hot flashes/flushes
Thyroid function, high (hyperthyroidism, thyrotoxicosis) (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Thyroid function, high (hyperthyroidism, thyrotoxicosis)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) — Diarrhea
Dysguesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Dysguesia
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Mucositis
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Nausea
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Vomiting
Hemorrhage, GU Vagina (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hemorrhage, GU Vagina
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Bacteremia
Blood infection - Ralstonia pickettii (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Blood infection - Ralstonia pickettii
Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infe (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection)(ANC <1.0 x 10e9/L, fever >=38.5 degrees C)
Infection with normal ANC or Grade 1 or 2 neutrophils Blood (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Infection with normal ANC or Grade 1 or 2 neutrophils Blood
Coagulase negative staph (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Coagulase negative staph
Infection with unknown ANC Oral cavity-gums (gingivitis) (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Thrush/candida
Infection with unknown ANC Upper airway NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Rhinovirus
Infection with unknown ANC Upper airway NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) — Infection with unknown ANC Upper airway NOS
Infection with unknown ANC Upper airway NOS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Rhinorrhea
Edema: limb (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Lower Extremity Edema
Lymphatics - Other (Fluid overload) (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Fluid overload
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) — Bilirubin (hyperbilirubinemia)
Creatinine (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) — Creatinine
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Hypokalemia
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Hypomagnesemia
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Hyponatremia
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Muscle weakness
Anxiety (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Anxiety
Depression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Depression
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Dizziness
Dry eye syndrome (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Dry eyes
Keratitis (corneal inflammation/corneal ulceration) (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Keratitis (corneal inflammation/corneal ulceration)
Pain Chest/thorax NOS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pain Chest/thorax NOS
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Headache
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Muscle pain
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Cough
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Shortness of breath
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) — Hypoxia
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Pleural effusion (non-malignant)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Corneal inflammation

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT00119366/Prot_SAP_000.pdf